CLINICAL TRIAL: NCT04026828
Title: Evaluation of Possible Genes in Periodontal Diseases by Genetic Methods
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Esra Guzeldemir-Akcakanat, Chair of the Department of Periodontology, Kocaeli University
Other Study IDs: KOU 2019/067
Record Dates: First submitted 2019-07-12; First posted 2019-07-19 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Generalized Aggressive Periodontitis; Chronic Periodontitis
Keywords: chronic periodontitis; aggressive periodontitis; expression; polymorphism; mutation
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gingival tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis Group: Chronic periodontitis and aggressive periodontitis patients
  Interventions: Genetic: Periodontitis Group
- Control Group: Both periodontal and medically healthy volunteers.
  Interventions: Genetic: Periodontitis Group

INTERVENTIONS:
Genetic: Periodontitis Group — Periodontitis group consists of both chronic and aggressive periodontitis patients

SUMMARY:
Generalized aggressive Periodontitis (GAgP) and chronic periodontitis (CP) are inflammatory diseases. Little is known about molecular changes and signaling cascade of host response. Inflammatory diseases are undercontrol of genetic and enviromental factors. Transcription factors are gene-specific factors that are often considered to act as a link connecting genetic and enviromental factors.

The aim of this study is to investigate the gene regions that are thought to play a role in the pathogenesis of GAgP and CP, and to interpret new and reliable pathognomonic-prognostic markers in the diagnosis and treatment of these diseases with the help of expression and mutation analyzes and polymorphism studies.

DETAILED DESCRIPTION:
Generalized aggressive Periodontitis (GAgP) is a multifactorial, destructive, inflammatory and complex disease. The progression of the disease is undercontrol of immunologic, microbiologic, environmental and genetic factors. The immunologic and genetic factors are not clearly defined yet.

Chronic periodontitis (CP) is an infectious disease resulting within the supporting tissues of the teeth. It is commonly detected in adults. CP is initiated and sustained by bacterial plaque.

Both AgP and CP are inflammatory diseases. Little is known about molecular changes and signaling cascade of host response. Inflammatory diseases are undercontrol of genetic and environmental factors. Transcription factors are gene-specific factors that are often considered to act as a link connecting genetic and environmental factors.

This research is a continuation project. In the previous 2 studies which were conducted and published with the support of TÜBİTAK 1001 and KOU BAP, it was found 2 gene regions thought to have an effect on GAgP and KP pathogenesis by genomics, proteomics and immunohistochemical methods; MZB1 and ECH1. The aim of this study is to confirm these gene regions by gene expression analysis, mutation analysis and polymorphism studies.

In the literature, there was no study on the genome analysis, protein activity and immunohistochemical examination of these genes in the CP and GAgP. There was no study that evaluated the expression, mutation and polymorphism studies.

The first 2 steps of the study were completed with the support provided by Kocaeli University Scientific Research Project Unit [119.500,00 TL (KOU BAP 2013/5)] and TUBITAK [(TÜBİTAK 1001 214S008, 261.500,00 TL)].

The aim of this study is to investigate the gene regions that are thought to play a role in the pathogenesis of GAgP and CP, and to interpret new and reliable pathognomonic-prognostic markers in the diagnosis and treatment of these diseases with the help of expression and mutation analyzes and polymorphism studies. Gene sites identified and clinically relevant in this study will serve as the basis for another study in which these genes are aimed at silencing.,,,

This research is a continuation project. In the previous 2 studies which were conducted and published with the support of TÜBİTAK 1001 and KOU BAP, it was found 2 gene regions that concluded which may have an effect on GAgP and KP pathogenesis by genomics, proteomics and immunohistochemical methods; MZB1 and ECH1. The aim of this study is to confirm these gene regions by gene expression analysis, mutation analysis and polymorphism studies.

ELIGIBILITY:
Inclusion criteria for aggressive periodontitis patients;

* The periodontal diagnosis of subjects with GAgP was established on the basis of clinical and radiographic criteria and was defined by the 1999 International World Workshop for a Classification of Periodontal Diseases and Conditions (Lang et al., 1999),
* Between 18 and 35 years of age,
* Otherwise healthy,
* The bone loss estimation was radiographically performed in each patient for the assessment of the extent and severity of alveolar bone loss.

Inclusion criteri for chronic periodontitis patients;

* Had at least 20 teeth,
* Exhibiting >30% of measured sites with 5mm clinical attachment loss,,
* Had bleeding on probing (BOP) at >50% of the proximal sites.

Inclusion criteri for control individuals;

- Overall healthy individuals (dental, periodontal and systemically)

Exclusion Criteria for all individuals;

* Had any known systemic diseases or conditions that can/could influence the periodontal status (cancer, cardiovascular and respiratory diseases),
* Any history of hepatitis and/or HIV infection,
* Immunosuppressive chemotherapy,
* Current pregnancy, planning a pregnancy or lactation,
* Requirement for antibiotic prophylaxis,
* Had oral diseases other than GAgP,
* Oongoing orthodontic therapy,
* A history of antibiotic therapy, or periodontal treatment within the preceding six months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Having aggressive or chronic periodontitis and healthy volenteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Quality and accuracy of the products of RNA and DNA | 6 months
  RNA and DNA will be isolated from cells and the quality and accuracy of the products will be tested by Agilent 2100 bioanalyzer chips and quatity of the products will be controlled by Nanodrop ND 1000 spectrophotometer.
Mutations Analysis | 6 Months
  Evaluation will be performed with DNA which extracted from tissues. Amplicons will be reproduced by multiplex PCR, analysed by Ion reporter and the outcomes will be evaluated with diverse online databases and clinical correlations.
Gene polymorphism | 6 Months
  Genes will evaluated by LightSNiPs

CONTACTS AND LOCATIONS:
Overall Officials: ESRA GUZELDEMIR-AKCAKANAT, DDS, PhD, Principal Investigator — Kocaeli University